CLINICAL TRIAL: NCT00148330
Title: An Open Label Extension of the Phase II/III Clinical Trial of Intravitreal Triamcinolone on the Effects and Safety of Clinically Significant Diabetic Macular Oedema That Persists After Laser Treatment
Brief Title: Open Label Extension of a Clinical Trial of Intravitreal Triamcinolone for Diabetic Macular Oedema-TDMX Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Sydney (Other)
Responsible Party: Professor Mark Gillies, Save Sight Institute, The University of Sudyney
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NHMRC project 402573
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2005-05

CONDITIONS: Diabetic Macular Oedema
Keywords: Diabetic macular oedema; Triamcinolone acetate; Intravitreal injection; Clinical trial; Laser treatment
MeSH Terms: interventions — Triamcinolone; Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Triamcinolone acetate — When indicated, intravitreal triamcinolone (0.1 ml of Kenacort 40© [40mg/ml triamcinolone acetonide, Bristol-Myers Squibb pharmaceuticals, Australia]) was injected into the vitreous under sterile conditions in a minor procedures area.
  Other Names: Kenacort 40©

SUMMARY:
This open label extension will treat all the eyes of study participants with active study medication (intravitreal triamcinolone) as well as standard laser treatment where appropriate.

The specific aims will be to test the following hypotheses:

* That intravitreal triamcinolone for diabetic macular oedema that persists or recurs after laser treatment remains efficacious over five years
* That intravitreal triamcinolone for diabetic macular oedema that persists or recurs after laser treatment retains a manageable and acceptable safety profile over five years

DETAILED DESCRIPTION:
A 25 fold increase in the risk of going blind on diagnosis of diabetes is one of the most daunting threats that patients face. People using insulin are particularly challenged because they are unable accurately to draw up their dose of drug. Most cases of vision impairment in diabetes are due to macular oedema that persists or recurs after laser treatment. There are now a number of uncontrolled, anecdotal reports that intravitreal triamcinolone (IVTA) is highly effective for the treatment of diabetic macular edema which is refractory to conventional laser treatment. We commenced the first placebo-controlled, double masked clinical trial of IVTA for refractory macular oedema in 2002. The 3 month results from this study provide the first scientific proof of principle that IVTA reduces macular thickness and improves vision. The two year results will be available in March 2005, but confidential interim analysis of efficacy data in September 2004 suggested that the beneficial effect of triamcinolone treatment persisted. Thus it appears that treatment with IVTA may be the most significant development for the prevention of blindness in people with diabetes since the introduction of laser treatment. It would also be a highly cost-effective intervention that could be administered by general ophthalmologists. The treatment cannot be recommended for routine use, however, until its long term efficacy and safety have been established. Since we already have a well studied group of patients who have received treatment for 2 years, we are in a unique position to extend the study in order to provide the long-term (5-year) safety and efficacy data that does not appear to be forthcoming from any other source. The completion of this study will have a direct and immediate effect on the risk of blindness in people with diabetes by allowing doctors to predict more accurately the long term effects of this promising new treatment.

ELIGIBILITY:
Inclusion Criteria:

Participation in the study will be offered to all patients at the conclusion of the TDMO study. Currently we are still following 64 of the 69 (93%) eyes that were initially entered into the study that had reduced vision from diabetic macular oedema at baseline.

Exclusion Criteria:

* Uncontrolled glaucoma
* Loss of vision due to other causes (e.g. age related macular degeneration, myopic macular degeneration)
* known allergies to triamcinolone acetate, patient is already receiving systemic steroid treatment, intercurrent severe disease such as septicemia, any condition which would affect follow-up or photographic documentation (e.g. geographical, psycho-social, media opacities)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2005-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Increase of ≥5 letters at the 5-year study visit on a LogMAR chart compared with (a) the initial baseline level and (b) the level at the 2-year study visit. | 3 year extension, total 5 years study from baseline
  Changes from Baseline to 5 years: Improvement of ≥5 letters after 5 years was found in 14/33 (42%) eyes initially treated with triamcinolone compared with 11/34 (32%) eyes initially treated with placebo (zGEE=0.81, P=0.4).
  Changes from 2 to 5 years (open-label extension):Improvement of ≥5 letters of best-corrected visual acuity was found in 8/29 (28%) eyes initial-triamcinolone compared with 7/28 (25%) initial-placebo eyes (zGEE=0.20, P=0.8).
Incidence of moderate or severe adverse events over the 3 years of the open-label extension | 3 year extension study, total 5 year study from baseline
  The incidence of cataract surgery declined in the third year: 5/11 (45%) eyes from the initial-triamcinolone group that were phakic at the beginning of the 3rd year required cataract surgery.

SECONDARY OUTCOMES:
Change in macular thickness by OCT | 3 year extension, total 5 year study from the baseline
  Changes from Baseline to 5 years: Foveal thickness had decreased by 30µm (95% confidence interval, -47 to 107µm) less in the initial-triamcinolone group than in the initial-placebo group at 5 years (zGEE=0.76, P=0.45).
  Changes from 2 to 5 years (open-label extension):Foveal thickness had actually increased slightly on average in the initial-triamcinolone group, but decreased in initial-placebo eyes. Overall it had decreased by 70µm (95% confidence interval, -1 to 140µm) more in the placebo group than in the treatment group between 2 and 5 years (zGEE=1.93, P=0.05).
Any change in visual acuity | 3 year extension, total 5 year study from the baseline
  Loss of ten or more letters was found in 6/33 (18%) initial-triamcinolone eyes compared with 8/34 (24%) initial-placebo eyes.
Number of laser treatments required. | 3 year extension study, total 5 year study from baseline
  During the third to fifth years of the study, a similar proportion of eyes from the 2 groups had macular edema that warranted laser treatment: initial-triamcinolone, 5/29 (17%); initial-placebo, 6/28 (21%).

CONTACTS AND LOCATIONS:
Overall Officials: Mark C Gillies, MBBS, PhD, Principal Investigator — Save Sight Institute, Deaprtment of Clinical Ophthalmology, University of Sydney
Locations (1):
- Save Sight Institute, Sydney/Sydney Eye Hospital Campus, University of Sydney, Sydney, New South Wales, Australia

REFERENCES:
- [Background] Sutter FK, Simpson JM, Gillies MC. Intravitreal triamcinolone for diabetic macular edema that persists after laser treatment: three-month efficacy and safety results of a prospective, randomized, double-masked, placebo-controlled clinical trial. Ophthalmology. 2004 Nov;111(11):2044-9. doi: 10.1016/j.ophtha.2004.05.025. PMID 15522370
- [Background] Larsson J, Zhu M, Sutter F, Gillies MC. Relation between reduction of foveal thickness and visual acuity in diabetic macular edema treated with intravitreal triamcinolone. Am J Ophthalmol. 2005 May;139(5):802-6. doi: 10.1016/j.ajo.2004.12.054. PMID 15860283
- [Background] Kuo CH, Gillies MC. Role of steroids in the treatment of diabetic macular edema. Int Ophthalmol Clin. 2009 Spring;49(2):121-34. doi: 10.1097/IIO.0b013e31819fcce8. No abstract available. PMID 19349792
- [Result] Gillies MC, Simpson JM, Gaston C, Hunt G, Ali H, Zhu M, Sutter F. Five-year results of a randomized trial with open-label extension of triamcinolone acetonide for refractory diabetic macular edema. Ophthalmology. 2009 Nov;116(11):2182-7. doi: 10.1016/j.ophtha.2009.04.049. Epub 2009 Oct 1. PMID 19796823
- [Result] Gillies M. Diabetic macular edema. Ophthalmology. 2009 Mar;116(3):595; author reply 596-7. doi: 10.1016/j.ophtha.2008.12.016. No abstract available. PMID 19264220
- [Result] Gillies MC, Simpson JM, Zhu M, Hunt G, Ali H, Gaston C. Intravitreal triamcinolone. Ophthalmology. 2009 Mar;116(3):591. doi: 10.1016/j.ophtha.2008.09.044. No abstract available. PMID 19264215
- [Result] Gillies MC, Sutter FK, Simpson JM, Larsson J, Ali H, Zhu M. Intravitreal triamcinolone for refractory diabetic macular edema: two-year results of a double-masked, placebo-controlled, randomized clinical trial. Ophthalmology. 2006 Sep;113(9):1533-8. doi: 10.1016/j.ophtha.2006.02.065. Epub 2006 Jul 7. PMID 16828501
- [Result] Larsson J, Kifley A, Zhu M, Wang JJ, Mitchell P, Sutter FK, Gillies MC. Rapid reduction of hard exudates in eyes with diabetic retinopathy after intravitreal triamcinolone: data from a randomized, placebo-controlled, clinical trial. Acta Ophthalmol. 2009 May;87(3):275-80. doi: 10.1111/j.1755-3768.2008.01245.x. Epub 2008 Sep 10. PMID 18785964
- [Derived] Wickremasinghe SS, Rogers SL, Gillies MC, Zhu M, Wong TY. Retinal vascular caliber changes after intravitreal triamcinolone treatment for diabetic macular edema. Invest Ophthalmol Vis Sci. 2008 Nov;49(11):4707-11. doi: 10.1167/iovs.08-1678. Epub 2008 Jul 3. PMID 18599569